CLINICAL TRIAL: NCT02236637
Title: A Prospective Registry of Patients With a Confirmed Diagnosis of Adenocarcinoma of the Prostate Presenting With Metastatic Castrate-Resistant Prostate Cancer
Brief Title: A Registry to Observe the Treatment of Prostate Cancer Under Routine Medical Care
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100857; 212082PCR4001 (Other: Janssen Pharmaceutica NV - CTMS ID)
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
Keywords: Adenocarcinoma of the Prostate; Registry; metastatic castration-resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mCRPC patients: Patients with metastatic castration-resistant prostate cancer treated according to routine clinical practice

SUMMARY:
The purpose of this registry is to document the characteristics and management of patients with metastatic castrate resistant prostate cancer (mCRPC) in routine clinical practice, independent of treatment used. Given the rapidly evolving landscape in mCRPC treatments, there is a need for a current and improved understanding of how these treatments fit into the current treatment paradigm for mCRPC, how they are combined and sequenced, and how their relative effectiveness profiles emerge outside of a clinical trial setting. This will be based on documentation and description of sequencing of treatment initiation, termination, and duration; relative effectiveness of treatments; defined medical resource utilization (MRU) and quality-of-life parameters and follow-up for survival.

DETAILED DESCRIPTION:
This is a non-interventional, multicenter, prospective registry of patients with a confirmed diagnosis of adenocarcinoma of the prostate presenting with mCRPC, based on documented metastatic prostate cancer and documented castration resistance. Castrate-resistant prostate cancer is defined by disease progression despite testosterone <50 ng/dL, and/or androgen deprivation therapy, and/or a history of orchiectomy, and may present as a continuous rise in prostate-specific antigen (PSA), and/or worsening of existing disease/symptoms, and/or the appearance of new metastases. Observational methodology will be used to capture data. The decision of patients to take part in the registry will not influence their medical care. Treatment decisions will be made at the discretion of the treating physician, per routine clinical practice. Only data available from routine clinical practice will be collected. It is expected that approximately 3,000 patients will participate in this registry. To ensure a patient population representative of clinical practice and to reduce selection bias, all patients meeting the eligibility criteria at a participating site should be consecutively enrolled in the registry, irrespective of their treatment. The planned total duration of the registry will be 5.5 years from the date that the first patient is enrolled, irrespective of the country or registry site. The anticipated duration of patient enrollment is 2.5 years. The maximum duration of follow-up for individual patients in the observational period of the registry will be 3 years, regardless of when they are enrolled. The 3-year period of the observational period will document the sequencing of systemic mCRPC treatments during routine clinical practice, considering the life expectancy of patients with mCRPC in the registry. Unless specified otherwise per local regulations, all patients must give their informed consent to participate in this registry before data collection (ie, data entry into the case report form [CRF]) is performed. Patients will be enrolled at the time of initiation of a new systemic mCRPC treatment or during a period when a patient is considered to be in surveillance according to clinical practice. Baseline data collection will include details of the patient's prostate cancer history and prior prostate cancer treatment. This will be followed by a prospective observational period during which patients may cycle through multiple systemic mCRPC treatment periods and periods of surveillance. During the observational period, data will be collected at the following time points of a patient's course of treatment in routine clinical practice: initiation of a new systemic mCRPC treatment; termination of a systemic mCRPC treatment; when the duration of a systemic mCRPC treatment or surveillance period is >3 months, data collection will be performed at a minimum frequency of 3-monthly intervals during that period. Survival data will be collected for all patients 3 years after their enrollment or at the close of the registry, whichever occurs first, except for those patients who withdraw their consent prior to completing the observation period.

ELIGIBILITY:
Inclusion Criteria:

Patients with a histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate Patients with documented metastatic prostate cancer Patients with documented castration resistance Patients either: Initiating a new systemic mCRPC treatment; or considered to be in surveillance according to clinical practice Sign (or their legally-acceptable representatives must sign) a participation agreement or informed consent form (ICF), per local regulations.

Exclusion Criteria:

Any patient who is withdrawn from the registry for any reason may not re-enter the registry

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 3,000 patients will be enrolled in this registry. Patients eligible for enrollment will be men aged at least 18 years, with a confirmed diagnosis of adenocarcinoma of the prostate, with documented metastatic prostate cancer and documented castration resistance. Patients will be enrolled at the time of initiating a new systemic anticancer mCRPC treatment or during surveillance; for the purpose of the registry, at enrollment, initiation of a new systemic mCRPC treatment is considered as ±30 days from a patient's baseline data collection.
Sampling Method: Probability Sample
Enrollment: 3050 (Actual)
Dates: Start 2013-06-14 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Sequencing of treatment initiation, termination, and duration | At baseline, at treatment initiation/termination and at least every 3 months during maximum 3 years
  During the registry all systemic mCRPC therapies, corticoids for systemic use in the context of prostate cancer treatment and local mCRPC therapies, including but not limited to urologic surgery, orthopaedic surgery, and local radiotherapy, will be documented.

SECONDARY OUTCOMES:
Clinical Benefit | At baseline, at treatment initiation/termination and at least every 3 months during maximum 3 years
  Clinical benefit will be based on the Eastern Cooperative Oncology Group (ECOG) performance status, which measure the patient status on a scale from 0 (fully active) to 5 (dead).
Medical Resource Utilization | At baseline, at treatment initiation/termination and at least every 3 months during maximum 3 years
  Total number of days of hospitalization due to prostate cancer, or treatment of the disease, total number of visits to an emergency room due to prostate cancer, or treatment of the disease, and total number of outpatient visits due to prostate cancer, or treatment of the disease
European Quality of Life-5 Dimensions, 5 Levels Questionnaire (EQ-5D-(5L)) | At baseline, at treatment initiation/termination and at least every 3 months during maximum 3 years
  The EQ-5D-5L is an instrument for measuring health status. It consists of the descriptive system and the EQ visual Analogue scale (EQ VAS). The descriptive system comprises the same 5 dimensions (mobility, self care, usual activities, pain/discomfort, and anxiety/depression). There are 5 levels for each dimension: no problems, slight problems, moderate problems, severe problems, and extreme problems. The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labeled 'the best health you can imagine' and 'the worst health you can imagine'.
Functional Assessment of Cancer Therapy - Prostate Cancer (FACT-P) | At baseline, at treatment initiation/termination and at least every 3 months during maximum 3 years
  The FACT-P consists of the FACT-General (FACT-G) and a prostate cancer subscale. The FACT-G (Version 4) contains a 27-item questionnaire and is composed of 4 subscales of health-related quality-of-life: physical well-being, social/family well-being, emotional well being, and functional well-being. The prostate cancer subscale is composed of 12 items, related to prostate-specific questions, which include sexuality, bowel/bladder function, and pain. The score for each of the 39 questions ranges from 0 to 4. The total FACT-P score thus ranges from 0 to 156; a higher score indicates better QOL
Overall Survival | At treatment initiation/termination or every 3 months from baseline to 3 years
Radiologic Assessment | At baseline, at treatment initiation/termination and at least every 3 months during maximum 3 years
  Radiologic assessment methodology and radiologic response will be documented. Prostate Cancer Working Group 2 (PCWG2) and Response Evaluation Criteria In Solid Tumor (RECIST) are recommended guidelines for assessment.
Prior prostate cancer treatment | At baseline
  Prior prostate cancer treatment (local and systemic therapy) from the time of diagnosis of prostate cancer to entry in the registry will be recorded.
Reason for start and rationale for choice of treatment | At treatment initiation during maximum 3 years
Reason for treatment discontinuation | At treatment discontinuation during maximum 3 years

CONTACTS AND LOCATIONS:
Locations (146):
- Austria (2):
  - Salzburg
  - Vienna
- Belgium (13):
  - Aalst
  - Antwerp
  - Bonheiden
  - Brasschaat
  - Bruges
  - Edegem
  - Ghent
  - Kortrijk
  - Liège
  - Ostend
  - Ottignies
  - Roeselare
  - Turnhout
- France (22):
  - Angers
  - Avignon
  - Béziers
  - Brest
  - Gap
  - Hyères
  - La Tronche
  - Marseille
  - Metz
  - Montpellier
  - Nancy
  - Paris
  - Périgueux
  - Pierre-Bénite
  - Pringy
  - Reims
  - Rennes
  - Saint-Grégoire
  - Saint-Mandé
  - Saint-Quentin
  - Toulouse
  - Tours
- Germany (25):
  - Augsburg
  - Bad Saarow
  - Bautzen
  - Berlin
  - Braunschweig
  - Chemnitz
  - Duisburg
  - Erkrath
  - Frankfurt
  - Hamburg
  - Holzminden
  - Jena
  - Kiel
  - Kirchheim
  - Nürtingen
  - Remscheid
  - Reutlingen
  - Rostock
  - Schwerin
  - Sindelfingen
  - Tübingen
  - Ulm
  - Weiden
  - Wilhelmshaven
  - Würselen
- Israel (5):
  - Beer Yaakov
  - Beersheba
  - Haifa
  - Holon
  - Tel Aviv
- Luxembourg (2):
  - Luxembourg
  - Niedercorn
- Poland (7):
  - Bydgoszcz
  - Gdynia
  - Krakow
  - Lodz
  - Opole
  - Poznañ
  - Warsaw
- Portugal (6):
  - Braga
  - Coimbra
  - Evora
  - Lisbon
  - Porto
  - Setúbal
- Russia (7):
  - Moscow
  - Obninsk
  - Omsk
  - Rostov-on-Don
  - Saint Petersburg
  - Ufa
  - Yekaterinburg
- Slovenia (3):
  - Celje
  - Ljubljana
  - Slovenj Gradec
- Spain (14):
  - A Coruña
  - Asturias
  - Barakaldo Vizcaya
  - Barcelona
  - Bilbao Vizcaya
  - Girona
  - Langreo
  - Palma de Mallorca
  - Pontevedra
  - Sabadell
  - Salamanca
  - Santiago de Compostela
  - Valladolid
  - Zaragoza
- Sweden (9):
  - Borås
  - Gothenburg
  - Malmo
  - Örebro
  - Östersund
  - Stockholm
  - Umeå
  - Vaxjo
  - Västerås
- Switzerland (2):
  - Aarau
  - Winterthur
- Turkey (Türkiye) (7):
  - Ankara
  - Edirne
  - Istanbul
  - Izmir
  - Kayseri
  - Kocaeli
  - Turkey
- United Kingdom (22):
  - Ashton-under-Lyne
  - Barnstaple
  - Blackburn
  - Bournemouth
  - Bradford
  - Brighton Sussex
  - Burton
  - Crewe
  - Huddersfield
  - Lancaster
  - Leeds Yorks
  - London
  - N/a N/a
  - Plymouth
  - Scunthorpe
  - Steeton
  - Stoke-on-Trent
  - Taunton
  - Torquay
  - Wakefield
  - Wigan
  - York

REFERENCES:
- [Derived] Verry C, Vincendeau S, Massetti M, Blachier M, Vimont A, Bazil ML, Bernardini P, Pettre S, Timsit MO. Pattern of Clinical Progression Until Metastatic Castration-Resistant Prostate Cancer: An Epidemiological Study from the European Prostate Cancer Registry. Target Oncol. 2022 Jul;17(4):441-451. doi: 10.1007/s11523-022-00899-6. Epub 2022 Jul 16. PMID 35841526
- [Derived] Bjartell A, Lumen N, Maroto P, Paiss T, Gomez-Veiga F, Birtle A, Kramer G, Kalinka E, Spaeth D, Feyerabend S, Matveev V, Lefresne F, Lukac M, Wapenaar R, Costa L, Chowdhury S. Real-World Safety and Efficacy Outcomes with Abiraterone Acetate Plus Prednisone or Prednisolone as the First- or Second-Line Treatment for Metastatic Castration-Resistant Prostate Cancer: Data from the Prostate Cancer Registry. Target Oncol. 2021 May;16(3):357-367. doi: 10.1007/s11523-021-00807-4. Epub 2021 Apr 7. PMID 33826036
- [Derived] Chowdhury S, Bjartell A, Lumen N, Maroto P, Paiss T, Gomez-Veiga F, Birtle A, Kramer G, Kalinka E, Spaeth D, Feyerabend S, Matveev V, Lefresne F, Lukac M, Wapenaar R, Costa L. Real-World Outcomes in First-Line Treatment of Metastatic Castration-Resistant Prostate Cancer: The Prostate Cancer Registry. Target Oncol. 2020 Jun;15(3):301-315. doi: 10.1007/s11523-020-00720-2. PMID 32500294